CLINICAL TRIAL: NCT03654456
Title: The Impact of Sleep Apnea on the Mortality of Sepsis - A Retrospective Study
Brief Title: Impact of Sleep Apnea on Sepsis Mortality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-06-019AC
Record Dates: First submitted 2018-07-24; First posted 2018-08-31 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Sleep Apnea Syndromes; Sepsis; Mortality
Keywords: obstructive sleep apnea; sepsis; outcome; prognosis; sleep-disordered breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Sepsis; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis patients with OSA: Sepsis patients who received a prior polysomnography showing an apnea-hypopnea index at least 5/hr with compatible symptoms
  Interventions: Biological: OSA
- Sepsis patients without OSA: Sepsis patients who received a prior polysomnography showing an apnea-hypopnea index less than 5/hr

INTERVENTIONS:
Biological: OSA — The diagnosis of OSA (obstructive sleep apnea) relies on polysomnographic data showing an apnea-hypopnea index at least 5/hr with compatible symptoms.
  Groups: Sepsis patients with OSA

SUMMARY:
By clinical record review, this retrospective study aims to compare the mortality of sepsis patients with versus without obstructive sleep apnea, who were diagnosed and treated in Taipei Veterans General Hospital, Taiwan.

DETAILED DESCRIPTION:
This retrospective study aims to compare the mortality of sepsis patients with versus without obstructive sleep apnea (OSA). Patients with a diagnosis of sepsis, who had received a prior polysomnography at Taipei Veterans General Hospital during Jan. 1, 2001 to May 31, 2017 will be enrolled. Obstructive sleep apnea (OSA) is defined by an apnea-hypopnea index at least 5/hr with compatible symptoms. Their clinical record will be reviewed and data including demography, polysomnography and details related to sepsis (source of infection, number of organ dysfunction at initial diagnosis of sepsis and survival time) will be collected. The start of the survival time (follow-up time) is the date when sepsis is diagnosed. The end of the survival time (follow-up time) is the date of death or end of hospitalization (date of discharge). Survival analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received received a polysomnography at Taipei Veterans General Hospital during Jan. 1, 2001 to May 31, 2017
2. Patients who were admitted with a diagnosis of sepsis after the polysomnography
3. The diagnosis of sepsis fulfilling the clinical criteria

Exclusion Criteria:

1. Younger than 20 years
2. Not compatible with a definition of sepsis
3. subjects with incomplete data

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sepsis Patients who had received a polysomnography at Taipei Veterans General Hospital during Jan. 1, 2001 to May 31, 2017 will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-05-27 (Estimated); Study Completion 2019-05-27 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 40 days
  percentage of sepsis patients died of sepsis

SECONDARY OUTCOMES:
Survival time | up to 40 days
  Survival time is defined as the length from the date when sepsis is diagnosed to date of discharge or death
Mortality | 7-day
  percentage of sepsis patients died of sepsis
Mortality | 28-day
  percentage of sepsis patients died of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ta Chou, M.D, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Result] Huang CY, Chen YT, Wu LA, Liu CJ, Chang SC, Perng DW, Chen YM, Chen TJ, Lee YC, Chou KT. Sleep apnoea patients have higher mortality when confronting sepsis. Eur J Clin Invest. 2014 Jan;44(1):38-45. doi: 10.1111/eci.12187. Epub 2013 Nov 11. PMID 24117403